CLINICAL TRIAL: NCT04155463
Title: Measurement of Agricultural and Dietary Glyphosate Exposure Among Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Cynthia Curl, Associate Professor, Boise State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K01ES028745 (NIH); K01ES028745 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Exposure to Herbicides
Keywords: Dietary Intervention; Glyphosate; Herbicide; Pregnancy; Agricultural Communities; Organic food

STUDY DESIGN:
Intervention Model Description: Study participants will take part in a two-week dietary intervention. All participants will receive one week of organic food and one week of conventional food, randomized to order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organic Diet, Then Conventional Diet: (Experimental): These participants first received an organic diet for one week. During that week, daily first morning void urine samples were collected. After a washout period of one day, these participants then received a conventional (non-organic) diet for one week. During that week, daily first morning void urine samples were collected.
  For each week, participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with either the organic diet or conventional diet. Study staff verified all food items corresponded with the dietary intervention that week, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
  Interventions: Other: Organic Diet; Other: Conventional Diet
- Conventional Diet, Then Organic Diet (Experimental): These participants first received a conventional (non-organic) diet for one week. During that week, daily first morning void urine samples were collected. After a washout period of one day, these participants then received an organic diet for one week. During that week, daily first morning void urine samples were collected.
  For each week, participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with either the organic diet or conventional diet. Study staff verified all food items corresponded with the dietary intervention that week, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
  Interventions: Other: Organic Diet; Other: Conventional Diet

INTERVENTIONS:
Other: Organic Diet — Participants receive one week of organic food. Organic food is certified through the USDA's National Organic Program as produced without the use of synthetic pesticides, including glyphosate.
Other: Conventional Diet — Participants receive one week of conventionally grown (non-organic) food.

SUMMARY:
The purpose of this research is to understand whether and how pregnant women may be exposed to glyphosate, the active ingredient in a common herbicide. The researchers aim to assess glyphosate exposure among pregnant women in Idaho, and to attribute that exposure to agricultural and dietary sources. Pregnant women who live either near or far from glyphosate-treated fields will be recruited for study inclusion, and exposure will be assessed via urinary biomonitoring on a weekly basis throughout pregnancy. Each participant will also take part in a two-week dietary intervention, during which they will receive one week of organic food and one week of conventional food, in a crossover design. Urinary biomonitoring will occur on a daily basis during the dietary intervention phase. The researchers hypothesize that women who live near agricultural fields treated with glyphosate will have higher exposures than those who live in non-agricultural regions, and that consumption of an organic diet will reduce exposures in both groups. All study components will be completed with no face-to-face interaction to eliminate all coronavirus (COVID-19) related risks.

DETAILED DESCRIPTION:
This study focuses on human exposure to glyphosate, the single most commonly applied agricultural chemical in the world. Glyphosate is an herbicide, and is most commonly known as the active ingredient in "Round Up". Glyphosate has been declared a probable human carcinogen by the International Agency for Research on Cancer and multiple toxicological studies have further suggested potential neurological and developmental effects of glyphosate exposure at environmentally-relevant levels. However, despite its extensive use, frequent presence in food and environmental media, and potential toxicity, current exposure levels in human populations are not well documented. This study aims to assess glyphosate exposure among a cohort of pregnant women and to quantify the relative contribution of agricultural and dietary sources of this exposure. A cohort of 40 pregnant women will be recruited from urban areas >10 miles from the nearest glyphosate-treated field and agricultural areas <1 mile from the nearest glyphosate-treated field. Weekly urine samples collected from these women throughout their pregnancies will be used to analyze glyphosate exposure. These same 40 participants will also take part in a two week-long randomized cross-over design dietary intervention, during which participants will receive one week of exclusively organic food (grown without the use of synthetic pesticides, including glyphosate) and one week of exclusively conventional food, in random order. During the intervention, the researchers will collect daily spot urine samples from each participant to analyze glyphosate exposure related to diet. The researchers hypothesize that during the time of year when glyphosate is actively applied, women living near glyphosate-treated fields will have higher exposures than those living further away. They also hypothesize that glyphosate exposure will be reduced among participants during randomization to the organic diet, but that this decrease will be larger among urban women than among those living near glyphosate-treated fields. The researchers have taken extra precautions to eliminate all COVID-specific risks. There will be no face-to-face contact between research staff and study participants throughout the entire study. Interactions between researchers and study participants will take place through videos, emails, texts, and/or phone calls. All urine samples will be left for researchers to pick up at a predetermined location and time, and all groceries will be delivered to participants' home and left at their front door.

ELIGIBILITY:
Inclusion Criteria:

* Be in the first trimester of pregnancy
* No diagnosis of gestational diabetes or other high risk pregnancy factors
* Consume an exclusively conventional diet with no intentions to switch to an organic diet
* Agree to refrain from applying residential glyphosate (Round Up) during the study
* Either live more than 10 miles or less than 1 mile from a glyphosate treated field

Exclusion Criteria:

- Occupational exposure to glyphosate, or live in a household with an individual with occupational glyphosate exposure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Curl, PhD, Principal Investigator — Boise State University
Locations (1):
- Boise State University, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 40 pregnant women in their first trimester from Women, Infants, and Children (WIC) clinics in Idaho as part of a longitudinal study to examine urinary glyphosate concentrations during pregnancy. We enrolled participants between February 23 and June 3, 2021 and followed them until they gave birth between August 5 and December 28, 2021. Of the 58 individuals referred by WIC clinics, 53 (91%) were eligible; 40 (75%) of eligible individuals were enrolled in the study.
Pre-assignment Details: As part of the longitudinal study, we conducted a two-week randomized crossover dietary intervention from June 16-June 30, 2021. 39 of the 40 participants took part in the dietary intervention (one participant was assigned to an arm but was out of town during the intervention). We randomly assigned participants to receive one week of either organic or conventional groceries, followed by one washout day, then one week of groceries of the opposite food type.
Period: First Intervention (1 Week)
Arm/Group | Organic Diet, Then Conventional Diet: | Conventional Diet, Then Organic Diet
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — out of town during dietary intervention | 0 | 1
Period: Washout (1 Day)
Arm/Group | Organic Diet, Then Conventional Diet: | Conventional Diet, Then Organic Diet
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Organic Diet, Then Conventional Diet: | Conventional Diet, Then Organic Diet
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Organic Diet, Then Conventional Diet:: These participants first received an organic diet for one week, defined as food certified through the United States Department of Agriculture's National Organic Program as produced without the use of synthetic pesticides, including glyphosate. During that week, daily first morning void urine samples were collected. After a washout period of one day, these participants then received a conventional (non-organic) diet for one week. During that week, daily first morning void urine samples were collected.
  For each week, participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with either the organic diet or conventional diet. Study staff verified all food items corresponded with the dietary intervention that week, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
- Conventional Diet, Then Organic Diet: These participants first received a conventional (non-organic) diet for one week. During that week, daily first morning void urine samples were collected. After a washout period of one day, these participants then received an organic diet for one week, defined as food certified through the United States Department of Agriculture National Organic Program as produced without the use of synthetic pesticides, including glyphosate.. During that week, daily first morning void urine samples were collected.
  For each week, participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with either the organic diet or conventional diet. Study staff verified all food items corresponded with the dietary intervention that week, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
- Total: Total of all reporting groups
Arm/Group | Organic Diet, Then Conventional Diet: | Conventional Diet, Then Organic Diet | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Customized [Count of Participants; unit: Participants]
  18-22 years | 6 | 5 | 11
  23-27 years | 4 | 6 | 10
  28-32 years | 6 | 7 | 13
  33-37 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could identify as more than one Race/Ethnicity
  Participants
    Caucasian or White | 9 | 11 | 20
    Hispanic or Latina | 10 | 9 | 19
    Asian | 1 | 0 | 1
    American Indian or Alaskan Native | 1 | 0 | 1
    African American or Black | 0 | 0 | 0
Highest Level of Education [Count of Participants; unit: Participants]
  Less than high school | 2 | 3 | 5
  Graduated high school/earned General Educational Development | 9 | 5 | 14
  Some college | 8 | 10 | 18
  Bachelor's degree | 1 | 0 | 1
  Graduate school/advanced degree | 0 | 1 | 1
Household income in previous year [Count of Participants; unit: Participants]
  < $10,000 - 19,999 | 5 | 4 | 9
  $20,000 - 29,999 | 3 | 7 | 10
  $30,000 - 30,999 | 3 | 5 | 8
  $40,000 - 59,999 | 4 | 1 | 5
  > $60,000 | 3 | 2 | 5
  Missing or prefer not to answer | 2 | 0 | 2
Number living in household [Count of Participants; unit: Participants]
  1-3 | 9 | 6 | 15
  4-6 | 10 | 12 | 22
  7-9 | 1 | 1 | 2
Personally used herbicides at residence in last year [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 20 | 19 | 39
Someone else used herbicides at residence in last year [Count of Participants; unit: Participants]
  Yes | 6 | 2 | 8
  No | 13 | 15 | 28
  Don't Know | 1 | 2 | 3
Type of herbicides used at residence in last year [Count of Participants; unit: Participants] — Population: This measure applies only to participants who indicated that they "Personally used herbicides at residence in last year" or "Someone else used herbicides at residence in last year" (i.e., this measure only applies to the 6 participants in the "Organic Diet, Then Conventional Diet" Arm and the 2 participants in the "Conventional Diet, Then Organic Diet" Arm that answered "Yes" to "Personally used herbicides at residence in last year" or "Someone else used herbicides at residence in last year.")
  Participants
    Don't know or unknown pesticides sprayed by pesticide control company: number analyzed (Participants) | 6 | 2 | 8
    Don't know or unknown pesticides sprayed by pesticide control company | 4 | 1 | 5
    Roundup® (glyphosate): number analyzed (Participants) | 6 | 2 | 8
    Roundup® (glyphosate) | 0 | 1 | 1
    Cheetah® (glufosinate ammonium): number analyzed (Participants) | 6 | 2 | 8
    Cheetah® (glufosinate ammonium) | 1 | 0 | 1
    Spectracide® (combination of non-glyphosate herbicides): number analyzed (Participants) | 6 | 2 | 8
    Spectracide® (combination of non-glyphosate herbicides) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Specific Gravity-adjusted Urinary Glyphosate Concentrations During Conventional and Organic Diet
Description: We collected 531 daily first morning void urine samples. We aliquoted 0.6 mL of each participant's seven daily urine samples to form a composite sample intended to represent each participant's mean glyphosate exposure during each week of the dietary intervention For all 39 participants there was one weekly composite urine sample from the conventional diet period and one weekly composite urine sample from the organic diet period. These 78 composite urine samples were analyzed for glyphosate concentrations and adjusted for urine specific gravity.
Time Frame: One week conventional diet and one week organic diet
Population: We geocoded each participant's address and verified the existence and location of all fields within a 0.5 km radius of their home. We report specific-gravity adjusted urinary glyphosate concentrations during the conventional and organic weeks for all participants and stratified by agricultural proximity, i.e. for participants living farther than 0.5 km of an agricultural field ("far-field") and living within 0.5 km of an agricultural field ("near-field").
Measure: Geometric Mean (Inter-Quartile Range); unit: ug/L
Units Other Than Participants: Composite Urine Samples
Groups:
- Conventional Diet: This arm refers to participants during their one week assigned to a conventional diet (regardless of whether they were assigned to receive conventional food the first week of the intervention or the second week of the intervention). During this time, participants received a conventional diet for one week. During that week, daily first morning void urine samples were collected.
  Participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with a conventional diet (i.e. no organic foods). Study staff verified all food items corresponded with a conventional diet, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
- Organic Diet: This arm refers to participants during their one week assigned to an organic diet (regardless of whether they were assigned to receive organic food the first week of the intervention or the second week of the intervention). During this time, participants received an organic diet for one week, defined as food certified through the United States Department of Agriculture National Organic Program as produced without the use of synthetic pesticides, including glyphosate. During that week, daily first morning void urine samples were collected.
  Participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with an organic diet. Study staff verified all food items corresponded with an organic diet, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
Arm/Group | Conventional Diet | Organic Diet
Number analyzed (Participants) | 39 | 39
Number analyzed (Composite Urine Samples) | 78 | 78
ug/L
  All Participants | 0.19 [0.11 to 0.30] | 0.17 [0.10 to 0.26]
  Far-field Participants: number analyzed (Participants) | 19 | 19
  Far-field Participants: number analyzed (Composite Urine Samples) | 38 | 38
  Far-field Participants | 0.18 [0.11 to 0.31] | 0.14 [0.10 to 0.23]
  Near-field Participants: number analyzed (Participants) | 20 | 20
  Near-field Participants: number analyzed (Composite Urine Samples) | 40 | 40
  Near-field Participants | 0.21 [0.12 to 0.29] | 0.20 [0.12 to 0.27]
Statistical Analysis 1: Comparison: Conventional Diet vs Organic Diet; Based on previous pesticide research, we calculated a sample size of 40 participants to provide a power of 0.80 at a 0.05 significance level in a two-sided test. We assumed a standard deviation of 0.5 µg/L; Test type: Other; p = 0.17, Wilcoxon signed rank test; Two-tailed test for paired data; Median Percent Change = -18.4 — This calculation shows the median percent change in urinary glyphosate concentrations going from the conventional diet to organic diet for all participants. Interquartile range for this was -37.4 to 29.8
Statistical Analysis 2: Comparison: Conventional Diet vs Organic Diet; Test type: Other; p = 0.06, Wilcoxon signed rank test; Two-tailed test for paired data; Median Percent Change = -24.2 — This calculation shows the median percent change in urinary glyphosate concentrations going from the conventional diet to organic diet for far-field participants. Interquartile range for this was -37.4 to -8.8
Statistical Analysis 3: Comparison: Conventional Diet vs Organic Diet; Test type: Other; p = 0.83, Wilcoxon (Mann-Whitney); Two-tailed test for paired data; Median Percent Change = 1.4 — This calculation shows the median percent change in urinary glyphosate concentrations going from the conventional diet to organic diet for near-field participants. Interquartile range for this was -41.9 to 43.0

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Organic Diet: This arm refers to all 39 participants during their one week assigned to an organic diet (regardless of whether they were assigned to receive organic food the first week of the intervention or the second week of the intervention). During this time, participants received an organic diet for one week, defined as food certified through the USDA's National Organic Program as produced without the use of synthetic pesticides, including glyphosate. During that week, daily first morning void urine samples were collected.
  Participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with an organic diet. Study staff verified all food items corresponded with an organic diet, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
- Conventional Diet: This arm refers to all 39 participants during their one week assigned to a conventional diet (regardless of whether they were assigned to receive conventional food the first week of the intervention or the second week of the intervention). During this time, participants received a conventional diet for one week. During that week, daily first morning void urine samples were collected.
  Participants ordered all food they anticipated eating that week (up to $150) from a unique account with a local grocery store in accordance with a conventional diet (i.e. no organic foods). Study staff verified all food items corresponded with a conventional diet, and then ordered the groceries to be delivered to the participant's home, when possible. For participants living in areas in which delivery was not available (generally rural areas), study staff picked up the food at the grocery store and delivered it to the participant's home.
Arm/Group | Organic Diet | Conventional Diet
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04155463/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04155463/SAP_002.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04155463/ICF_000.pdf